CLINICAL TRIAL: NCT00352365
Title: A Phase II Study of Lenalidomide (REVLIMID, NSC-703813) for Previously Untreated Non-M3, Deletion 5q Acute Myeloid Leukemia (AML) in Patients Age 60 or Older Who Decline Remission Induction Chemotherapy
Brief Title: Lenalidomide in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00785; NCI-2009-00785 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S0605; CDR0000484449; S0605 (Other: Southwest Oncology Group); S0605 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Lenalidomide

ARMS (1):
- Treatment (lenalidomide) (Experimental): INDUCTION THERAPY: Patients receive oral lenalidomide once daily on days 1-14, 1-21, or 1-28 (course 1). Patients undergo bone marrow biopsy on day 28 or 35 to assess treatment efficacy. Patients with stable or improving disease (i.e., a decrease in blast percentage) without progressive disease proceed to maintenance therapy.
  MAINTENANCE THERAPY: Beginning within 42 days after completion of induction therapy, patients receive oral lenalidomide once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid

SUMMARY:
This phase II trial is studying how well lenalidomide works in treating older patients with acute myeloid leukemia with abnormal chromosome 5q. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test whether the complete response rate among older patients with previously untreated acute myeloid leukemia (AML) with the del (5q) cytogenetic abnormality treated with lenalidomide is sufficiently high to warrant a phase III investigation.

II. Estimate the frequency and severity of toxicities of this drug in these patients.

III. Correlate, in a preliminary manner, additional cytogenetic abnormalities with response to lenalidomide.

IV. Estimate the total (complete and partial) response rate and the cytogenetic response rate in these patients.

OUTLINE:

INDUCTION THERAPY: Patients receive oral lenalidomide once daily on days 1-14, 1-21, or 1-28 (course 1). Patients undergo bone marrow biopsy on day 28 or 35 to assess treatment efficacy. Patients with stable or improving disease (i.e., a decrease in blast percentage) without progressive disease proceed to maintenance therapy.

MAINTENANCE THERAPY: Beginning within 42 days after completion of induction therapy, patients receive oral lenalidomide once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Morphologically confirmed diagnosis of acute myeloid leukemia (AML) by bone marrow aspiration and biopsy within the past 14 days

  * Diagnostic biopsy within the past 28 days with marrow blast percentage ≥ 70% allowed provided no potentially antileukemic therapy was received after biopsy
* Cytogenetic evidence of del (5q) abnormality by conventional karyotyping or fluorescence in situ hybridization (FISH)
* Previously untreated disease

  * Must have declined standard AML cytotoxic chemotherapy regimens
* WBC ≤ 30,000/mm³
* History of prior myelodysplastic syndromes (MDS) allowed
* No acute promyelocytic leukemia (FAB M3)
* No blastic transformation of chronic myelogenous leukemia
* Zubrod performance status 0-2
* Bilirubin ≤ 2.5 times upper limit of normal (ULN) (unless elevation is due primarily to elevated unconjugated hyperbilirubinemia secondary to Gilbert's syndrome or hemolysis, but not to liver dysfunction)
* AST and ALT ≤ 3.5 times ULN
* Creatinine ≤ 1.5 times ULN
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception at least 4 weeks prior to, during, and for 4 weeks after completion of study treatment
* No known allergy to thalidomide
* Concurrent enrollment on SWOG-S9910 allowed (for SWOG patients)
* No prior systemic chemotherapy for acute leukemia except hydroxyurea

  * Single-dose intrathecal chemotherapy allowed before or concurrently with induction chemotherapy
* No prior AML induction-type chemotherapy or high-dose chemotherapy with hematopoietic stem cell support
* Prior hematopoietic growth factors, thalidomide, arsenic trioxide, signal-transduction inhibitors, azacitidine, and low-dose cytarabine (i.e., < 100 mg/m²/day) for treatment of MDS allowed
* At least 30 days since prior therapy for MDS (excluding growth factors)
* No prior lenalidomide for MDS
* At least 6 months since prior chemotherapy or radiotherapy for another malignancy
* No concurrent therapy for another malignancy
* Concurrent hormonal therapy allowed

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-06; Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikkael Sekeres, Principal Investigator — SWOG Cancer Research Network
Locations (54):
- United States (54):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Shasta Regional Medical Center, Redding, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Salina Regional Health Center, Salina, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison Bremerton Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Oncology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Sekeres MA, Gundacker H, Lancet J, Advani A, Petersdorf S, Liesveld J, Mulford D, Norwood T, Willman CL, Appelbaum FR, List AF. A phase 2 study of lenalidomide monotherapy in patients with deletion 5q acute myeloid leukemia: Southwest Oncology Group Study S0605. Blood. 2011 Jul 21;118(3):523-8. doi: 10.1182/blood-2011-02-337303. Epub 2011 May 6. PMID 21551228

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide: Induction Therapy: Oral lenalidomide once daily on days 1-14, 1-21, or 1-28. Maintenance Therapy: Oral lenalidomide once daily on days 1-21 (1 cycle = 28 days)
Period: Induction Therapy
Arm/Group | Lenalidomide
Started | 41
Eligible | 38
Eligible and Began Protocol Therapy | 37
Completed | 14
Not Completed | 27
Not completed — Adverse Event | 7
Not completed — Progression/Relapse | 8
Not completed — Death | 7
Not completed — Not protocol specified | 1
Not completed — Not eligible | 3
Not completed — Death before starting protocol therapy | 1
Period: Maintenance Therapy
Arm/Group | Lenalidomide
Started | 12
Eligible and Began Protocol Therapy | 8
Completed | 0
Not Completed | 12
Not completed — Progression/Relapse | 3
Not completed — Death | 2
Not completed — Not protocol specified | 3
Not completed — Not eligible | 4

BASELINE CHARACTERISTICS:
Population: Eligible patients who began protocol therapy
Groups:
- Induction Therapy: Oral lenalidomide once daily on days 1-14, 1-21, or 1-28
Arm/Group | Induction Therapy
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 73.7 [60.1 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3
  White | 33
  Unknown or Not Reported | 1
Hispanic [Number; unit: participants]
  Yes | 1
  No | 32
  Unknown | 4
Disease Onset [Number; unit: participants]
  De Novo | 16
  Treatment related | 2
  MDS related | 19
Performance Status [Number; unit: participants] — Performance status is graded according to the Zubrod Performance Status Scale. Patients with a performance status of 0 are fully active, able to carry on all pre-disease performance without restriction. Patients with a performance status of 1 are restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  participants
    0 | 7
    1 | 30

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 5 years
Population: Eligible patients who received any treatment and were assessed for toxicity were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- Maintenance Therapy: Oral lenalidomide once daily on days 1-21 (1 cycle = 28 days)
Arm/Group | Induction Therapy | Maintenance Therapy
Number analyzed (Participants) | 37 | 8
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1 | 0
  AST, SGOT | 1 | 0
  Adult respiratory distress syndrome (ARDS) | 1 | 0
  Anorexia | 1 | 0
  Bilirubin (hyperbilirubinemia) | 1 | 0
  Calcium, serum-low (hypocalcemia) | 3 | 0
  Cardiac-ischemia/infarction | 1 | 0
  Cough | 1 | 0
  Creatinine | 3 | 0
  Dermatology/Skin-Other (Specify) | 1 | 0
  Diarrhea | 2 | 0
  Dyspnea (shortness of breath) | 2 | 0
  Fatigue (asthenia, lethargy, malaise) | 11 | 0
  Febrile neutropenia | 15 | 2
  Glucose, serum-high (hyperglycemia) | 2 | 0
  Hemoglobin | 7 | 2
  Induration/fibrosis (skin and subcutaneous tissue) | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Esophagus | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lip/perioral | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 5 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 0 | 1
  Leukocytes (total WBC) | 14 | 4
  Lymphopenia | 2 | 0
  Muscle weakness, not d/t neuropathy - body/general | 3 | 0
  Nausea | 1 | 0
  Neuropathy: motor | 1 | 0
  Neutrophils/granulocytes (ANC/AGC) | 16 | 5
  Platelets | 21 | 3
  Pneumonitis/pulmonary infiltrates | 4 | 0
  Potassium, serum-low (hypokalemia) | 3 | 0
  Pulmonary/Upper Respiratory-Other (Specify) | 2 | 0
  Rash/desquamation | 2 | 0
  Renal failure | 1 | 0
  Sodium, serum-high (hypernatremia) | 1 | 0
  Sodium, serum-low (hyponatremia) | 1 | 1
  Vomiting | 1 | 0

2. Secondary Outcome: Cytogenetic Abnormalities
Description: Number of baseline cytogenetic abnormalities by responders (CR, CRi, and PR) and nonresponders.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: Number of abnormalities
Groups:
- Responders: Eligible and evaluable patients who achieved CR/CRi/PR
- Nonresponders: Eligible and evaluable patients who did not achieve CR/CRi/PR
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 5 | 32
Number of abnormalities | 8 [1 to 20] | 8 [0 to 31]

3. Secondary Outcome: Total Response
Description: Morphologic complete remission (CR): ANC >=1,000/mcl, platelet count >=100,000/mcl, <5% bone marrow blasts, no Auer rods, no evidence of extramedullary disease. Morphologic complete remission with incomplete blood count recovery (CRi): Same as CR but ANC may be <1,000/mcl and/or platelet count <100,000/mcl. Partial remission (PR): ANC >1,000/mcl, platelet count >100,000/mcl, and at least 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts <5% with persistent Auer rods.
Time Frame: Up to 5 years
Population: Eligible patients who began protocol therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Therapy
Number analyzed (Participants) | 37
percentage of participants | 14 [5 to 29]

4. Primary Outcome: Complete Response
Description: Morphologic complete remission (CR): ANC >=1,000/mcl, platelet count >=100,000/mcl, <5% bone marrow blasts, no Auer rods, no evidence of extramedullary disease. Morphologic complete remission with incomplete blood count recovery (CRi): Same as CR but ANC may be <1,000/mcl and/or platelet count <100,000/mcl.
Time Frame: Up to 5 years
Population: Eligible patients who began protocol therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Therapy
Number analyzed (Participants) | 37
percentage of participants | 11 [3 to 25]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Induction Therapy | Maintenance Therapy
Serious Adverse Events (participants affected / at risk) | 24/37 | 4/8
Other Adverse Events (participants affected / at risk) | 34/37 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Therapy (N=37) | Maintenance Therapy (N=8)
Blood/Bone Marrow-Other (Specify) (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 2
Hemoglobin (Blood and lymphatic system disorders) | 2 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI - Colon (Gastrointestinal disorders) | 0 | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Esophagus (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 3 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 1 | 0
Infection with unknown ANC - Blood (Infections and infestations) | 1 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 | 0
AST, SGOT (Investigations) | 1 | 0
Leukocytes (total WBC) (Investigations) | 0 | 1
Lymphopenia (Investigations) | 1 | 0
Platelets (Investigations) | 3 | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 1
Pain - Head/headache (Nervous system disorders) | 1 | 0
Syncope (fainting) (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Therapy (N=37) | Maintenance Therapy (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 0
Hemoglobin (Blood and lymphatic system disorders) | 23 | 5
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 8 | 2
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 7 | 1
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 0 | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Edema: limb (General disorders) | 9 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 18 | 5
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 3 | 1
Pain - Pain NOS (General disorders) | 2 | 0
Rigors/chills (General disorders) | 4 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 5 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4 | 0
AST, SGOT (Investigations) | 6 | 1
Alkaline phosphatase (Investigations) | 2 | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 9 | 1
Creatinine (Investigations) | 8 | 1
Leukocytes (total WBC) (Investigations) | 20 | 5
Lymphopenia (Investigations) | 2 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 20 | 5
Platelets (Investigations) | 24 | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8 | 2
Anorexia (Metabolism and nutrition disorders) | 6 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 11 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 15 | 2
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7 | 1
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Neuropathy: motor (Nervous system disorders) | 2 | 0
Neuropathy: sensory (Nervous system disorders) | 4 | 0
Pain - Head/headache (Nervous system disorders) | 3 | 1
Taste alteration (dysgeusia) (Nervous system disorders) | 2 | 1
Mood alteration - anxiety (Psychiatric disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae/purpura (hemorrhage into skin or mucosa) (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 7 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 | 2
Hematoma (Vascular disorders) | 0 | 1
Hot flashes/flushes (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less